CLINICAL TRIAL: NCT05879341
Title: The Effect of Irisin Polymorphism on Cognitive Function and Inter-individual Exercise Response Variability
Brief Title: Effect of Gene Polymorphism on Cognitive Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Dean-Chuan Wang, PhD, Associate Professor, Kaohsiung Medical University Chung-Ho Memorial Hospital
Other Study IDs: KMUHIRB-G(I)-20220005
Record Dates: First submitted 2023-04-06; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Polymorphosis; Cognitive Function
Keywords: Irisin; Cognition; Polymorphism; High intensity interval training
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample will be collected from the participants which will be used to extract serum and DNA. Serum will be used to measure Irisin and BDNF levels.
  DNA will be used for BDNF and Irisin SNP Geno-typing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: High intensitiy interval training — The participants will perform HIIT at 85% of their heart rate reserve. There will be 8 cycles of high intensity with four minutes of rest intervals in between.
  Other Names: HIIT; High intensity interval Exercise

SUMMARY:
The goal of this observational study is to study the effect of gene polymorphism on cognitive improvement in response to exercise in healthy participants. The main questions it aims to answer are:

To investigate whether FNDC5/Irisin genotype polymorphism affects cognitive function and inter-individual variability in exercise response.

To explore whether the FNDC5/Irisin gene polymorphism can act alone or interact with the BDNF gene to cause inter-individual differences in cognitive function responses to exercise gain.

Participants will be asked to perform high-intensity interval training( HIIT) on a cycle ergometer. Each high-intensity training period will be 30 seconds followed by a 4-minute rest period.

The participants will also perform cognitive tests (Vistorian stroop test and Fitlight trainer test) before and after the exercise.

DETAILED DESCRIPTION:
Exercise has a significant effect on improving brain function. It can improve cognitive function, enhance learning effects, and prevent the occurrence of neurodegenerative diseases in the elderly. Exercise's mechanism of action to improve cognitive function includes stimulating the nervous system to secrete brain-derived neurotrophic factor (BDNF) and skeletal muscle to secrete irisin. However, the effect of exercise on improving physical function varies from person to person. This phenomenon is called inter-individual exercise response variability. Genetic differences may be responsible for this phenomenon. The genotype differences of BDNF and Irisin can cause cognitive function. However, the scientific community is still unclear whether the differences between the two genotypes are related to individual differences in exercise responses. The investigators suspect that genotype might be responsible for interindividual variability in motor responses and therefore designed this experiment to test this thesis. This study is expected to recruit 200 healthy adults to complete the genotype sequencing of BDNF and Irisin and use the cognitive function responses before and after a single high-intensity interval aerobic exercise to establish the model that genotype affects the variability of individual exercise responses. The experimental results of this study can help the scientific community understand the influence of genotype on individual differences in exercise response and further explore and refine the design of exercise prescription.

ELIGIBILITY:
Inclusion Criteria:

* Taiwanese National who perform less than 120 minutes of aerobic exercise per week.

The subjects will refrain from drinking alcoholic or caffeinated drinks 24 hours prior to the participation in the study

Exclusion Criteria:

Subjects who are diagnosed with

* Hypertension
* Arrhythmia
* Depression
* Color blindness
* Musculoskeletal injury within one year

Body Mass index higher than 25

Pregnant females

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Taiwanese National who perform less than 120 minutes of aerobic exercise per week.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change in Serum BDNF levels | The blood sample will be collected immediately after the participant has signed the consent to assess pre exercise BDNF levels
  Serum brain derived neurotrophic factor levels
Change in Serum BDNF levels | The blood sample will be collected 30 minutes after the participant has completed high intensity exercise to assess post exercise BDNF levels
  Serum brain derived neurotrophic factor levels
Change in Serum Irisin Levels | The blood sample will be collected immediately after the participant has signed the consent to assess pre exercise Irisin levels
  Serum Irisin levels
Change in Serum Irisin Levels | The blood sample will be collected 30 minutes after the participant has completed high intensity exercise to assess post exercise Irisin levels
  Serum Irisin levels
Change in Stroop Reaction time | Baseline
  Reaction time for Victorian version of Stroop test
Change in Stroop Reaction time | Immediately after the procedure
  Reaction time for Victorian version of Stroop test
Change in Fitlight reaction time | Baseline
  Mean Reaction time to Fitlight Trainer complex patterns
Change in Fitlight reaction time | Immediately after the procedure
  Mean Reaction time to Fitlight Trainer complex patterns

SECONDARY OUTCOMES:
Monitor the Heart rate | During the procedure
  Effect of gene polymorphism on changes in heart rate variability due to exercise.
Change in Fitlight simple reaction time | Baseline
  Reaction time to Fitlight
Change in Fitlight simple reaction time | Immediately after the procedure
  Reaction time to Fitlight

CONTACTS AND LOCATIONS:
Overall Officials: Dean-Chuan Wang, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No